CLINICAL TRIAL: NCT01024166
Title: A Usability Study of Patient-Reported Outcomes (PRO)-Based Palliative and Hospice Care Practice: Integrating PROs and Decision Support Into an Electronic Record
Brief Title: Patient-Reported Outcomes-Based Palliative and Hospice Care Practice: A Usability Study
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2009-0776
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Advanced Cancers
Keywords: Cancer; Patient-Reported Outcomes Computer System; PRO; Palliative Care; Symptoms; Questionnaire; Patients; Caregivers; Palliative Care Physicians; Palliative Care Nurses
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patient: Patient computer system use questionnaire
  Interventions: Behavioral: Questionnaire and Review Session
- Caregiver: Caregiver computer system use questionnaire
  Interventions: Behavioral: Questionnaire and Review Session
- Healthcare Provider: Physician and Nurse computer system use questionnaire
  Interventions: Behavioral: Questionnaire and Review Session

INTERVENTIONS:
Behavioral: Questionnaire and Review Session — Use PRO computer system to complete 2 questionnaires about any symptoms patient may be experiencing and their overall health, 30 minutes to complete. Review session about use of computer system and suggested changes.
  Other Names: Survey; Computer Program
  Groups: Caregiver; Patient
Behavioral: Questionnaire and Review Session — Use PRO computer system to complete 4 questionnaires about symptoms their overall health of patients, 30 minutes to complete. Review session about use of computer system and suggested changes.
  Other Names: Survey; Computer Program
  Groups: Healthcare Provider

SUMMARY:
The goal of this research study is to learn if palliative care patients or caregivers, and palliative care physicians or nurses can use a computer program designed to provide information about the symptoms and overall health of cancer patients.

DETAILED DESCRIPTION:
The Patient-Reported Outcomes (PRO) Computer System:

The PRO computer system used in this study has been designed to help doctors and nurses check the symptoms and overall health status of patients with cancer by reviewing the computer entries of patients and caregivers. The system has also been designed to help doctors and nurses make decisions about how to care for patients based on the computer entries.

Questionnaire and Review Session:

If you agree to take part in this study, you will have an questionnaire and review session at the Palliative Care outpatient clinic. The session will be conducted by a research staff member, but the study chair and/or other study staff members may also attend the session. The questionnaire and review session will have 3 steps, which are described below:

* If you are a patient receiving palliative care, you will use the PRO computer system to complete 2 questionnaires about any symptoms you may be experiencing and your overall health. If you are a caregiver for someone who is receiving palliative care, you will use the PRO computer system to complete 2 questionnaires about any symptoms that the patient you are caring for may be experiencing and their overall health. The study staff will instruct you on how to use the PRO computer system.
* If you are a physician or nurse, you will use the PRO computer system to complete 4 questionnaires about the symptoms and overall health of patients who are receiving palliative care. The study staff will instruct you on how to use the PRO computer system.
* You will then look at the results of the questionnaires you have completed, which will be shown to you in both number and graph form. You will also be shown other features and potential uses of the PRO computer system.
* Last, you will be asked about how easily you were able to use the computer system. You will also be asked about any changes you think could make the program easier to use.

The questionnaire and review session should take about 30 minutes to complete.

Study Data:

Your responses to the questionnaires will be destroyed after the questionnaire and review session. The responses you give when asked about the use of the PRO computer system will be kept after the questionnaire and review session. Only the study staff will have access to your responses. However, your responses will be coded with a study ID number, not by your name. Your saved responses will be stored in password-protected files that are available only to the study staff for 3 years.

Length of Study:

Your participation in this study will be over after you complete the questionnaire and review session.

This is an investigational study.

Up to 9 patients and 9 caregivers will take part in this study. All will be enrolled at M. D. Anderson.

Up to 9 physicians and nurses (4-5 of each) will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All patient/caregiver participants will be adults 21 years of age or older.
2. Participants will be palliative care cancer patients and/or their designated caregivers.
3. Participating patients should be receiving palliative care at the MD Anderson Cancer Center as an inpatient or have attended at least one outpatient appointment; participating caregivers should have provided care to their patient during an inpatient stay or have attended at least one outpatient appointment with their patient.
4. Physicians and nurses who are experts in palliative care will be eligible for study participation. For this study's purposes, a physician or nurse with a minimum of four years of experience working in a palliative care setting will be considered an expert in palliative care.

Exclusion Criteria:

1. Patients or caregivers who are not able to report on symptom status using the electronic measurement system.
2. Patient, caregivers, physicians, or nurses who do not agree to sign the study's informed consent documents.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Palliative care patients receiving care at University of Texas MD Anderson Cancer Center and their caregivers, physicians and nurses, all over the age of 21.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2009-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of System Usability of the Prototype Solution (Questionnaire Responses) | Single assessment point

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Kallen, PhD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org